CLINICAL TRIAL: NCT04726553
Title: Nature of Anifrolumab Impact on Vaccine-Emergent Immunity in Patients With Moderately to Severely Active Systemic Lupus Erythematosus: A Multi-Centre Open Label Parallel Group Trial:
Brief Title: Nature of Anifrolumab Impact on Vaccine-Emergent Immunity in SLE
Acronym: NAIVE
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oklahoma Medical Research Foundation (Other)
Collaborators: NYU Langone Health (Other); Yale University (Other); Piedmont Heart Institute, Inc., Atlanta, GA (Industry); Columbia University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D3461C00023; IRB 20-27 (Other: OMRF)
Record Dates: First submitted 2021-01-22; First posted 2021-01-27 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Systemic Lupus Erythematosus (SLE)
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — anifrolumab; Standard of Care; Azathioprine; Methotrexate; Mycophenolic Acid; Adrenal Cortex Hormones; Antimalarials

STUDY DESIGN:
Intervention Model Description: Parallel Groups will include ten SLE patients who receive anifrolumab added to standard of care and ten patients who receive only standard of care
Masking Description: There will be no masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Anifrolumab plus Standard of Care (Experimental): Anifrolumab will be added to Standard of Care Treatments for SLE
  Interventions: Drug: Anifrolumab
- Standard of Care (Placebo Comparator): Standard of Care Treatments for SLE
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Anifrolumab — Anifrolumab is a monoclonal antibody which inhibits the Interferon alpha beta receptor (IFNAR) which is the main transducer of signals from Type I interferons.
  Other Names: Medi 546
  Arms: Anifrolumab plus Standard of Care
Drug: Standard of Care — Standard of Care treatments for Systemic Lupus Erythematosus
  Other Names: azathioprine, methotrexate, mycophenolate mofetil, corticosteroids, antimalarials
  Arms: Standard of Care

SUMMARY:
This study to examines the impact of anifrolumab on disease activity, immune phenotypes, and development of neutralizing antibodies to quadrivalent influenza vaccine in patients with Systemic Lupus Erythematosus (SLE). 10 patients with moderately to severely active SLE will be treated with anifrolumab in addition to standard of care lupus treatments and 10 will receive only standard of care medications. All will receive influenza vaccine.

DETAILED DESCRIPTION:
This group of researchers previously observed that lupus patients with an elevated interferon alpha signal produced less neutralizing antibody to influenza vaccine which was directly or indirectly associated with increased flares and autoantibody production after immunization. Anifrolumab is an inhibitor of signaling through the Type I interferon alpha beta receptor. The current study is an open label parallel group pilot study to examine the impact of anifrolumab on development of neutralizing antibodies to quadrivalent influenza vaccine in patients with SLE. 10 patients with moderately to severely active SLE will initiate treatment with anifrolumab while continuing standard of care medications and 10 will receive only standard of care medications. Two weeks after baseline all will receive influenza vaccine. Blood samples will be drawn at baseline (Day 0), just prior to immunization (Week 2), and Weeks 4, 8, 12 and 16. Disease activity, gene/cytokine expression, autoantibody production and patient reported outcomes will also be tracked.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures.
2. Female and/or male aged 18 to 70 years inclusive.
3. Meet the 2019 European League Against Rheumatism/American College of Rheumatology Classification Criteria for Systemic Lupus.
4. Have moderate to severely active signs or symptoms defined as an SLE Disease Activity Index (SLEDAI) score of at least 6 or at least one moderately to severely active manifestation scoring B or A on British Isles Lupus Assessment Group (BILAG) Index.
5. May be taking up to 30 mg oral prednisone daily (or equivalent steroid) that has been stable for ≥ two weeks at the Baseline Visit.
6. May be taking antimalarial treatment at any tolerated dose that has been stable for ≥ two months at the Baseline Visit.

7, May be taking one oral or injectable standard of care immunosuppressant defined as: Any of the following medications administered for a minimum of 12 weeks prior to signing the informed consent, and at a stable dose for a minimum of 8 weeks prior to signing the informed consent through Day 0: (i) Azathioprine ≤200 mg/day (ii) Antimalarial (eg, chloroquine, hydroxychloroquine, quinacrine) (iii) Mycophenolate mofetil ≤2 g/day or mycophenolic acid ≤1.44 g/day (iv) Oral, subcutaneous (SC), or intramuscular methotrexate ≤25 mg/week

8. Non steroidal anti-inflammatory drugs (NSAIDS), topical or ocular steroids, or topical or ocular calcineurin inhibitors are allowed with any dosing schedule (prn or fixed dosing).

9. Female subjects must use 2 effective methods of avoiding pregnancy, only one of which is a barrier method, from the time they sign consent until 12 weeks after the last dose of study medication unless the subject is surgically sterile (e.g. bilateral oophorectomy or complete hysterectomy), has a sterile male partner, is at least 1 year postmenopausal, or practices sustained abstinence consistent with the subject's customary lifestyle. Postmenopausal is defined as at least 1 year since last menses and the subject has an elevated follicle-stimulating hormone (FSH) level greater than the threshold laboratory value of post-menopausal at screening. Effective methods of birth control include those listed in Appendix 12.8. Ineffective methods that should not be used are listed in Appendix 12.9

10. All males (sterilized or non-sterilized) who are sexually active must use condom (with spermicide where commercially available for contraception) from Day 1 until at least 12 weeks after receipt of the final dose of IP. It is strongly recommended that the female partner of a male subject also use an effective method of contraception from Appendix 12,8 in the protocol (other than a barrier method) throughout this period. Male subjects must not donate sperm during the course of the study and for 12 weeks after the last dose of the investigational product.

11. Females with an intact cervix must have documentation of a normal Pap smear with no documented malignancy or abnormalities (e.g., cervical intraepithelial neoplasia grade III, carcinoma in situ, or adenocarcinoma in situ within 2 years prior to randomization. Any abnormal Pap smear result documented within 2 years prior to randomization must be repeated to confirm patient eligibility.

12. Meets all of the following tuberculosis criteria:

* No signs or symptoms of active tuberculosis prior to or during Screening.
* No medical history suggestive of active tuberculosis.
* No recent contact with a person with active tuberculosis OR if there has been such contact, referral to a physician specializing in tuberculosis to undergo additional evaluation prior to randomization (documented comprehensively in source), and, if warranted, receipt of appropriate treatment for latent tuberculosis at or before the first administration of investigational product.
* No history of latent tuberculosis prior to initial Screening visit, with the exception of latent tuberculosis with documented completion of appropriate treatment.

  13. Testing for Inclusion in the Study for those in the anifrolumab arm:

Purified Protein Derivative or Tuberculosis spot test within 12 weeks prior to or during screening; if negative, subject is eligible. If positive or indeterminate, subject must undergo repeat test and chest x-ray. If both negative, subject is eligible.

Coronavirus disease (COVID-19) negative polymerase chain reaction test or equivalent test for active infection such as rapid antigen test result during screening period and no known or suspected exposure within 2 weeks prior to screening. If there is a known or suspected exposure, a subject must be negative upon retest obtained 2 weeks after exposure and must remain asymptomatic for inclusion in the study.

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to all staff at the Coordinating Clinic and/or at the study site)
2. Have already received the 2020-2021 quadrivalent influenza vaccine.
3. Receipt of any of the following:

   Any live or attenuated vaccine within 8 weeks prior to signing the ICF. Administration of killed vaccines is acceptable as long as not the influenza vaccine.

   Bacillus Calmette-Guerin (BCG) vaccine within 1 year of signing the ICF

   Blood transfusion or receipt of blood products within 4 weeks prior to signing the informed consent form (ICF)
4. For patients with active or ongoing nephritis there must be two proteinuria data points available within the last two months to confirm a stable protein/creatine ratio as defined by no increase of > 400 mg/gm between the first and second collection. There may be a delay of up to two weeks between screening and baseline for a repeat protein/creatinine ratio to be performed. The criteria will apply to the most recent two tests.
5. In the opinion of the investigator, the patient has any active, unstable organ-threatening manifestations of SLE. At the investigator's discretion there may be a delay of up to two weeks between screening and baseline for appropriate diagnostic testing to confirm this criterion is not met.
6. Lactating or pregnant females or females who intend to become pregnant or begin breastfeeding anytime from initiation of Screening until the end of the 12-week safety follow-up period following last dose of IP.
7. Spontaneous or induced abortion, still or live birth, or pregnancy ≤4 weeks prior to signing the informed consent form (ICF).
8. History of cancer, apart from:

   Squamous or basal cell carcinoma of the skin treated with documented success of curative therapy ≥3 months prior to Week 0 (Day 1).

   Cervical cancer in situ treated with apparent success with curative therapy ≥1 year prior to Week 0 (Day 1).
9. Recent infection requiring hospitalization or use of intravenous anti-infectives within four weeks of signing the informed consent form or oral anti-infectives within two weeks of baseline or known history of splenectomy.
10. Any elevation in liver function tests within two months prior to signing the informed consent or at the Screening visit will require reflex screening for active hepatitis. Any confirmed positive screening for hepatitis serology will be exclusionary including:

    1. Hepatitis B surface antigen (HBsAg), OR
    2. Hepatitis B core antibody (HBcAb) AND hepatitis B virus (HBV) DNA detected above the lower limit of quantitation (LLOQ) by reflex testing by the central laboratory at screening.
    3. Positive test for hepatitis C antibody as confirmed by central laboratory.
11. Other infections:

    1. Any clinical cytomegalovirus (CMV) or Epstein-Barr virus infection that has not completely resolved within 12 weeks prior to signing the ICF.
    2. Opportunistic infection requiring hospitalization or IV antimicrobial treatment within 3 years of randomization.
    3. Clinically significant chronic infection (e.g., osteomyelitis, bronchiectasis, etc) within 8 weeks prior to signing the informed consent form (ICF) (chronic nail infections are allowed).
12. For subjects to receive anifrolumab: any severe case of herpes zoster infection at any time prior to Baseline, including, but not limited to, non-cutaneous herpes (ever), herpes encephalitis (ever), recurrent herpes zoster (defined as 2 episodes within 2 years) or ophthalmic herpes involving the retina (ever). Any herpes zoster infection that has not completely resolved within 12 weeks prior to signing the ICF. History of positive hepatitis C antibody, hepatitis B virus surface antigen or hepatitis B virus core antibody.
13. Liver function tests (AST/ALT) > 2.5 X upper limit of normal for the testing laboratory for any cause.
14. Urine dipstick >/= 2+ with reflex protein/creatinine ratio >/= 3 gm/gm
15. White blood cells </= 2.0 x 10,9 Hg </= 7.0 mg/dl, or platelets dropping from normal values to </= 100 x 109 unless stable for two assessments at least one week apart or any platelet counts </=40 x 109 even if stable.
16. Known to have tested positive for human immunodeficiency virus.
17. Any history of severe COVID-19 infection (e.g. requiring hospitalization, intensive care unit (ICU) care or assisted ventilation) or any prior COVID-19 infection with unresolved sequelae.
18. Participation in another clinical study in which an investigational product that is not currently marketed was received during the last two months prior to Screening or for five half-lives of that study agent, whichever is longer.
19. Currently receiving any medications restricted by this protocol within two months or five half-lives of the agent whichever is longer: to include any cytotoxic agent (e.g. cyclophosphamide) or a marketed biologic agent (e.g. belimumab, abatacept, infliximab, any Tumor Necrosis Factor inhibitor, or any of the agents listed in the Appendix 12.11 of the protocol).
20. Persistent toxicities as per Common Terminology Criteria for Adverse Events (CTCAE) that is > grade 2 and caused by current treatments.
21. Hypersensitivity including anaphylaxis, known history of allergy or reaction to any component of the investigational product (IP) formulation or history of anaphylaxis to any human gamma globulin therapy (anifrolumab group only)
22. Known history of drug or alcohol abuse considered clinically significant by the investigator within one year of screening
23. Major surgery within 8 weeks before signing the informed consent form (ICF) or elective major surgery planned during the study period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in immune response to quadrivalent flu vaccine | 6 weeks after vaccination (8 weeks after baseline)
  Combined endpoint incorporating percentile ranks of log10 transformed ratios of antibody concentration and results of a hemagglutination inhibition assay.

SECONDARY OUTCOMES:
Proportion of patients who develop changes in autoantibodies after immunization with quadrivalent flu vaccine | 6 weeks after vaccination (8 weeks after baseline)
  Change will be defined as two-fold increase in titre, two-fold decrease, or new appearance at any titre
Proportion of patients who develop flares after immunization with quadrivalent flu vaccine | 6 weeks after vaccination (8 weeks after baseline)
  Flares will be defined as moderate or severe flares measured by modified SLEDAI Flare Index

CONTACTS AND LOCATIONS:
Overall Officials: Joan T Merrill, M.D., Study Director — Member; Cristina Arriens, M.D., Principal Investigator — Clinical Assistant Member
Locations (5):
- United States (5):
  - Yale University Medical Center, New Haven, Connecticut
  - Piedmont Hospital, Atlanta, Georgia
  - New York University Medical Center, New York, New York
  - Columbia Unversity Medical Center, New York, New York
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: Yes
de-identified data will be made available for sharing with other researchers upon application to our registry and approval by the internal review board of the Oklahoma Medical Research Foundation
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: one year after completion of the study
Access Criteria: Our registry requires registry board approval and internal review board approval. Investigators may apply with a description of the planned project

REFERENCES:
- [Background] Crowe SR, Merrill JT, Vista ES, Dedeke AB, Thompson DM, Stewart S, Guthridge JM, Niewold TB, Franek BS, Air GM, Thompson LF, James JA. Influenza vaccination responses in human systemic lupus erythematosus: impact of clinical and demographic features. Arthritis Rheum. 2011 Aug;63(8):2396-406. doi: 10.1002/art.30388. PMID 21598235
- [Background] Battafarano DF, Battafarano NJ, Larsen L, Dyer PD, Older SA, Muehlbauer S, Hoyt A, Lima J, Goodman D, Lieberman M, Enzenauer RJ. Antigen-specific antibody responses in lupus patients following immunization. Arthritis Rheum. 1998 Oct;41(10):1828-34. doi: 10.1002/1529-0131(199810)41:103.0.CO;2-T. PMID 9778224
- [Background] Abu-Shakra M, Press J, Buskila D, Sukenik S. Influenza vaccination of patients with systemic lupus erythematosus: safety and immunogenecity issues. Autoimmun Rev. 2007 Sep;6(8):543-6. doi: 10.1016/j.autrev.2006.12.004. Epub 2007 Jan 9. PMID 17854746
- See also: this is the institutional website of the sponsor. Ongoing research projects and further references can be found on that site — http://www.omrf.org